CLINICAL TRIAL: NCT00877929
Title: An 8-week Randomised, Double-blind Study to Compare the Fixed-dose Combination of Telmisartan 80 + Amlodipine 10mg Versus Amlodipine 10 mg Monotherapy as First Line Therapy in Type 2 Diabetes Patients With Hypertension.
Brief Title: Telmisartan Fixed Dose Combination vs Amlodipine in Hypertensive Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1235.21; 2008-000874-19 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-02-06; First posted 2009-04-08 (Estimated); Results first posted 2011-06-07 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

ARMS (2):
- Telmisartan 80 / Amlodipine 10 (Experimental): Telmisartan 80 / Amlodipine 5 for two weeks, then forced titration to Telmisartan 80 / Amlodipine 10 Fixed Dose Combination
  Interventions: Drug: Telmisartan 80; Drug: Amlodipine 10
- Amlodipine 10 (Active Comparator): Amlodipine 5 for two weeks, then forced titration to Amlodipine 10
  Interventions: Drug: Amlodipine 10

INTERVENTIONS:
Drug: Telmisartan 80 — Telmisartan 80 mg
  Arms: Telmisartan 80 / Amlodipine 10
Drug: Amlodipine 10 — Amlodipine 5 for two weeks, then forced titration to Amlodipine 10
  Arms: Telmisartan 80 / Amlodipine 10
Drug: Amlodipine 10 — Amlodipine 5 for two weeks, then forced titration to Amlodipine 10
  Arms: Amlodipine 10

SUMMARY:
To demonstrate that the fixed dose combination of telmisartan and amlodipine is more effective in lowering blood pressure.

ELIGIBILITY:
Inclusion criteria:

1. Hypertension defined as a mean in-clinic seated cuff Systolic Blood Pressure >150 mmHg at Visit 3 (Randomisation visit)
2. Diagnosis of Type 2 diabetes mellitus
3. =18 years of age at the date of signing the informed consent
4. Ability to stop current antihypertensive therapy without unacceptable risk to the patient (investigator's discretion)
5. Ability to provide written informed consent

Exclusion criteria:

1. Pre-menopausal women (last menstruation <=1 year prior to start of run-in period) who:

   1. are not surgically sterile; and/or
   2. are nursing or pregnant, or
   3. are of child-bearing potential and are NOT practicing acceptable means of birth control or do NOT plan to continue practising an acceptable method throughout the study.

   The only acceptable methods of birth control are:
   * Intrauterine device (IUD);
   * Oral contraceptives (started at least three months prior to start of run-in period)
   * Implantable or injectable contraceptives and
   * Estrogen patch
2. Night shift workers who routinely sleep during the daytime and whose work hours include midnight to 4:00 a.m.
3. Known or suspected secondary hypertension (e.g., renal artery stenosis, phaeochromocytoma)
4. Mean seated Systolic Blood Pressure (SBP) =180 mm Hg and/or mean seated Diastolic Blood Pressure (DBP) =110 mm Hg during any visit of the screening and placebo run-in periods
5. Patients with Type 1 diabetes mellitus
6. Renal dysfunction as defined by the following laboratory parameters: Serum creatinine >3.0 mg/dL (or >265 µmol /L) or known creatinine clearance <30 mL/min or clinical markers of severe renal impairment
7. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post-renal transplant patients or patients with only one kidney
8. Clinically relevant hypokalaemia or hyperkalaemia
9. Uncorrected sodium or volume depletion
10. Primary aldosteronism
11. Hereditary fructose intolerance
12. Biliary obstructive disorders (e.g., cholestatis) or hepatic insufficiency
13. Congestive heart failure New York Heart Academy (NYHA) functional class CHF III-IV (Refer to Appendix 10.3)
14. Contraindication to a placebo run-in period (e.g., stroke with-in the past six months, myocardial infarction, cardiac surgery, percutaneous transluminal coronary angioplasty, unstable angina or coronary artery bypass graft within the past three months prior to start of run-in period)
15. Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the Investigator
16. Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
17. Patients whose diabetes has not been stable and controlled for at least the past three months as defined by an HbA1C >10%
18. Patients who have previously experienced symptoms characteristic of angioedema during treatment with Angiotensin Converting Enzyme (ACE) inhibitors or angiotensin-II receptor antagonists
19. History of drug or alcohol dependency within six months prior to signing the informed consent form
20. Concomitant administration of any medications known to affect blood pressure, except medications allowed by the protocol
21. Any investigational drug therapy within one month of signing the informed consent
22. Known hypersensitivity to any component of the study drugs (telmisartan, amlodipine, or placebo)
23. History of non-compliance or inability to comply with prescribed medications or protocol procedures
24. Any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of telmisartan and amlodipine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (65):
- United States (15):
  - 1235.21.901 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1235.21.907 Boehringer Ingelheim Investigational Site, Tustin, California
  - 1235.21.913 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1235.21.910 Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - 1235.21.903 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1235.21.905 Boehringer Ingelheim Investigational Site, Tucker, Georgia
  - 1235.21.916 Boehringer Ingelheim Investigational Site, Olive Branch, Mississippi
  - 1235.21.915 Boehringer Ingelheim Investigational Site, Hickory, North Carolina
  - 1235.21.906 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1235.21.902 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1235.21.904 Boehringer Ingelheim Investigational Site, Penndel, Pennsylvania
  - 1235.21.908 Boehringer Ingelheim Investigational Site, Carrollton, Texas
  - 1235.21.909 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1235.21.912 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1235.21.911 Boehringer Ingelheim Investigational Site, Ettrick, Virginia
- Argentina (5):
  - 1235.21.102 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1235.21.103 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1235.21.107 Boehringer Ingelheim Investigational Site, Ramos Mejía
  - 1235.21.101 Boehringer Ingelheim Investigational Site, Santa Fe
  - 1235.21.105 Boehringer Ingelheim Investigational Site, Zárate
- Mexico (6):
  - 1235.21.302 Boehringer Ingelheim Investigational Site, Acapulco
  - 1235.21.304 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 1235.21.301 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1235.21.303 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1235.21.305 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1235.21.306 Boehringer Ingelheim Investigational Site, Guadalajara
- Netherlands (9):
  - 1235.21.408 Boehringer Ingelheim Investigational Site, Beek en Donk
  - 1235.21.401 Boehringer Ingelheim Investigational Site, Hoogwoud
  - 1235.21.405 Boehringer Ingelheim Investigational Site, Musselkanaal
  - 1235.21.404 Boehringer Ingelheim Investigational Site, Nijverdal
  - 1235.21.403 Boehringer Ingelheim Investigational Site, Oude Pekela
  - 1235.21.409 Boehringer Ingelheim Investigational Site, Roelofarensveen
  - 1235.21.406 Boehringer Ingelheim Investigational Site, The Hague
  - 1235.21.407 Boehringer Ingelheim Investigational Site, Voerendaal
  - 1235.21.402 Boehringer Ingelheim Investigational Site, Wildervank
- Slovakia (9):
  - 1235.21.501 Boehringer Ingelheim Investigational Site, Bratislava
  - 1235.21.502 Boehringer Ingelheim Investigational Site, Bratislava
  - 1235.21.503 Boehringer Ingelheim Investigational Site, Bratislava
  - 1235.21.504 Boehringer Ingelheim Investigational Site, Bratislava
  - 1235.21.507 Boehringer Ingelheim Investigational Site, Dunajská Streda
  - 1235.21.509 Boehringer Ingelheim Investigational Site, Martin
  - 1235.21.505 Boehringer Ingelheim Investigational Site, Nitra
  - 1235.21.506 Boehringer Ingelheim Investigational Site, Nitra
  - 1235.21.508 Boehringer Ingelheim Investigational Site, Rimavská Sobota
- South Africa (7):
  - 1235.21.27005 Boehringer Ingelheim Investigational Site, Cape Town
  - 1235.21.27007 Boehringer Ingelheim Investigational Site, Cape Town
  - 1235.21.27004 Boehringer Ingelheim Investigational Site, Durban
  - 1235.21.27006 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1235.21.27002 Boehringer Ingelheim Investigational Site, Krugersdorp
  - 1235.21.27001 Boehringer Ingelheim Investigational Site, Lenasia
  - 1235.21.27003 Boehringer Ingelheim Investigational Site, Pretoria
- South Korea (5):
  - 1235.21.202 Boehringer Ingelheim Investigational Site, Incheon
  - 1235.21.201 Boehringer Ingelheim Investigational Site, Seoul
  - 1235.21.203 Boehringer Ingelheim Investigational Site, Seoul
  - 1235.21.204 Boehringer Ingelheim Investigational Site, Seoul
  - 1235.21.205 Boehringer Ingelheim Investigational Site, Seoul
- Spain (5):
  - 1235.21.702 Boehringer Ingelheim Investigational Site, Castellon
  - 1235.21.705 Boehringer Ingelheim Investigational Site, Centelles
  - 1235.21.703 Boehringer Ingelheim Investigational Site, Sant Adrià Del Besós
  - 1235.21.704 Boehringer Ingelheim Investigational Site, Santa Coloma de Gramanet (Barcelona)
  - 1235.21.706 Boehringer Ingelheim Investigational Site, Santa Coloma de Gramanet
- Sweden (4):
  - 1235.21.801 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1235.21.803 Boehringer Ingelheim Investigational Site, Helsingborg
  - 1235.21.804 Boehringer Ingelheim Investigational Site, Lund
  - 1235.21.802 Boehringer Ingelheim Investigational Site, Västerås

RESULTS

PARTICIPANT FLOW:
Groups:
- Telmisartan 80 mg + Amlodipine 10 mg: Once daily Telmisartan 80 mg (T80) / Amlodipine 5 mg (A5) tablet for first 2 weeks then Telmisartan 80 mg (T80) / Amlodipine 10 mg (A10) tablet for 6 weeks.
- Amlodipine 10 mg: Once daily Placebo / Amlodipine 5 mg (A5) tablet for first 2 weeks then Placebo / Amlodipine 10 mg (A10) tablet for 6 weeks.
Period: Overall Study
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Started | 352 | 354
Completed | 332 | 319
Not Completed | 20 | 35
Not completed — Adverse Event | 11 | 20
Not completed — Protocol Violation | 3 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lack of Efficacy | 0 | 1
Not completed — Other reason (not specified) | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg | Total
Number analyzed (Participants) | 352 | 354 | 706
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (10.4) | 60.5 (9.7) | 60.5 (10.1)
Age, Customized [Number; unit: participants]
  < 65 years | 214 | 235 | 449
  >= 65 years | 138 | 119 | 257
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 169 | 341
  Male | 180 | 185 | 365
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian/Alaska Native | 7 | 5 | 12
  Asian | 30 | 40 | 70
  Black/African American | 43 | 41 | 84
  Hawaiian/Pacific Islander | 2 | 0 | 2
  White | 270 | 268 | 538
Region of Enrollment [Number; unit: participants]
  Spain | 19 | 18 | 37
  Mexico | 27 | 29 | 56
  Netherlands | 44 | 42 | 86
  Argentina | 33 | 31 | 64
  Republic of Korea | 9 | 11 | 20
  Sweden | 11 | 10 | 21
  Slovakia | 36 | 40 | 76
  United States | 120 | 121 | 241
  South Africa | 53 | 52 | 105
Race class [Number; unit: participants]
  Non-black | 309 | 313 | 622
  Black | 43 | 41 | 84
Height [Mean (Standard Deviation); unit: centimeter] | 167.1 (10.3) | 167.6 (10.9) | 167.4 (10.6)
Weight [Mean (Standard Deviation); unit: kilogram] | 90.2 (20.9) | 89.5 (19.4) | 89.9 (20.2)
Body Mass Index [Mean (Standard Deviation); unit: kilogram / square meter] | 32.1 (6.0) | 31.8 (6.1) | 32.0 (6.1)
Body Mass Index Class [Number; unit: participants]
  < 25 kg/square meter | 32 | 31 | 63
  25 to <30 kg/square meter | 114 | 123 | 237
  >= 30 kg/square meter | 206 | 200 | 406
Smoking history [Number; unit: participants]
  Never smoked | 221 | 222 | 443
  Ex-smoker | 91 | 89 | 180
  Currently smokes | 40 | 43 | 83
Alcohol history [Number; unit: participants]
  Non drinker | 227 | 218 | 445
  Drinks - no interference | 125 | 136 | 261

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure to Week 8
Description: Trough blood pressure measurements were the measurements observed at the end of the dosing interval just prior to the next dose of medication.
Time Frame: Baseline, week 8
Population: Treated Set includes all randomized participants who took at least one dose of treatment
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 320 | 311
mmHg | -29.0 (0.66) | -22.9 (0.67)
Statistical Analysis 1: Comparison: Telmisartan 80 mg + Amlodipine 10 mg vs Amlodipine 10 mg; Test type: Superiority or Other; p = 0.0001, ANCOVA; Included effects of treatment, week and treatment-by-week interaction with covariate of baseline blood pressure and baseline-week interaction; Mean Difference (Final Values) = -6.1, 95% CI [-7.9 to -4.2]

2. Secondary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure to Week 6
Description: as for outcome 1
Time Frame: Baseline, week 6
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 326 | 317
mmHg | -29.7 (0.62) | -22.6 (0.63)
Statistical Analysis 1: Comparison: Telmisartan 80 mg + Amlodipine 10 mg vs Amlodipine 10 mg; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.1, 95% CI [-8.9 to -5.4]

3. Secondary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure to Week 4
Description: as for outcome 1
Time Frame: Baseline, week 4
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 329 | 326
mmHg | -27.7 (0.62) | -21.1 (0.62)
Statistical Analysis 1: Comparison: Telmisartan 80 mg + Amlodipine 10 mg vs Amlodipine 10 mg; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.6, 95% CI [-8.3 to -4.9]

4. Secondary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure to Week 2
Description: as for outcome 1
Time Frame: Baseline, week 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 333 | 332
mmHg | -22.4 (0.65) | -16.4 (0.65)
Statistical Analysis 1: Comparison: Telmisartan 80 mg + Amlodipine 5 mg vs Amlodipine 5 mg; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.1, 95% CI [-7.9 to -4.3]

5. Secondary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure to Week 1
Description: as for outcome 1
Time Frame: Baseline, week 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 334 | 336
mmHg | -17.5 (0.61) | -12.6 (0.61)
Statistical Analysis 1: Comparison: Telmisartan 80 mg + Amlodipine 5 mg vs Amlodipine 5 mg; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.9, 95% CI [-6.6 to -3.2]

6. Secondary Outcome: Blood Pressure (BP) Control (SBP<140 mmHg, DBP<90 mmHg) at Eight Weeks
Description: Mean seated SBP<140 mmHg and mean seated DBP<90 mmHg
Time Frame: Baseline, week 8
Population: Treated set using last observation carried forward (LOCF)
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 329
participants | 237 | 177

7. Secondary Outcome: BP Control (SBP<140 mmHg, DBP<90 mmHg) at Six Weeks
Description: Mean seated SBP<140 mmHg and mean seated DBP<90 mmHg
Time Frame: Baseline, week 6
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 328
participants | 245 | 168

8. Secondary Outcome: BP Control (SBP<140 mmHg, DBP<90 mmHg) at Four Weeks
Description: Mean seated SBP<140 mmHg and mean seated DBP<90 mmHg
Time Frame: Baseline, week 4
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 329 | 326
participants | 235 | 155

9. Secondary Outcome: BP Control (SBP<140 mmHg, DBP<90 mmHg) at Two Weeks
Description: Mean seated SBP<140 mmHg and mean seated DBP<90 mmHg
Time Frame: Baseline, week 2
Population: Treated set using LOCF
Measure: Number; unit: participants
Groups:
- Telmisartan 80 mg + Amlodipine 5 mg: Once daily Telmisartan 80 mg (T80) / Amlodipine 5 mg (A5) tablet for first 2 weeks then Telmisartan 80 mg (T80) / Amlodipine 10 mg (A10) tablet for 6 weeks.
- Amlodipine 5 mg: Once daily Placebo / Amlodipine 5 mg (A5) tablet for first 2 weeks then Placebo / Amlodipine 10 mg (A10) tablet for 6 weeks.
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 337 | 341
participants | 184 | 103

10. Secondary Outcome: BP Control (SBP<140 mmHg, DBP<90 mmHg) at One Week
Description: Mean seated SBP<140 mmHg and mean seated DBP<90 mmHg
Time Frame: Baseline, week 1
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 334 | 336
participants | 130 | 72

11. Secondary Outcome: BP Control (SBP<130 mmHg, DBP<80 mmHg) at Eight Weeks
Description: Mean seated SBP<130 mmHg and mean seated DBP<80 mmHg
Time Frame: Baseline, week 8
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 329
participants | 121 | 59

12. Secondary Outcome: BP Control (SBP<130 mmHg, DBP<80 mmHg) at Six Weeks
Description: Mean seated SBP<130 mmHg and mean seated DBP<80 mmHg
Time Frame: Baseline, week 6
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 328
participants | 134 | 60

13. Secondary Outcome: BP Control (SBP<130 mmHg, DBP<80 mmHg) at Four Weeks
Description: Mean seated SBP<130 mmHg and mean seated DBP<80 mmHg
Time Frame: Baseline, week 4
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 329 | 326
participants | 94 | 38

14. Secondary Outcome: BP Control (SBP<130 mmHg, DBP<80 mmHg) at Two Weeks
Description: Mean seated SBP<130 mmHg and mean seated DBP<80 mmHg
Time Frame: Baseline, week 2
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 337 | 341
participants | 58 | 23

15. Secondary Outcome: BP Control (SBP<130 mmHg, DBP<80 mmHg) at One Week
Description: Mean seated SBP<130 mmHg and mean seated DBP<80 mmHg
Time Frame: Baseline, week 1
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 334 | 336
participants | 35 | 12

16. Secondary Outcome: Systolic Blood Pressure (SBP) Control 140 at Eight Weeks
Description: Mean seated SBP < 140 mmHg
Time Frame: Baseline, week 8
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 329
participants | 243 | 187

17. Secondary Outcome: SBP Control 140 at Six Weeks
Description: Mean seated SBP < 140 mmHg
Time Frame: Baseline, week 6
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 328
participants | 251 | 177

18. Secondary Outcome: SBP Control 140 at Four Weeks
Description: Mean seated SBP < 140 mmHg
Time Frame: Baseline, week 4
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 329 | 326
participants | 243 | 163

19. Secondary Outcome: SBP Control 140 at Two Weeks
Description: Mean seated SBP < 140 mmHg
Time Frame: Baseline, week 2
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 337 | 341
participants | 193 | 112

20. Secondary Outcome: SBP Control 140 at One Week
Description: Mean seated SBP < 140 mmHg
Time Frame: Baseline, week 1
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 334 | 336
participants | 141 | 81

21. Secondary Outcome: SBP Control 130 at Eight Weeks
Description: Mean seated SBP < 130 mmHg
Time Frame: Baseline, week 8
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 329
participants | 157 | 89

22. Secondary Outcome: SBP Control 130 at Six Weeks
Description: Mean seated SBP < 130 mmHg
Time Frame: Baseline, week 6
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 328
participants | 164 | 81

23. Secondary Outcome: SBP Control 130 at Four Weeks
Description: Mean seated SBP < 130 mmHg
Time Frame: Baseline, week 4
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 329 | 326
participants | 137 | 70

24. Secondary Outcome: SBP Control 130 at Two Weeks
Description: Mean seated SBP < 130 mmHg
Time Frame: Baseline, week 2
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 337 | 341
participants | 92 | 42

25. Secondary Outcome: SBP Control 130 at One Week
Description: Mean seated SBP < 130 mmHg
Time Frame: Baseline, week 1
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 334 | 336
participants | 50 | 26

26. Secondary Outcome: SBP Response 140 at Eight Weeks
Description: SBP < 140 mmHg or a reduction >=10 mmHg
Time Frame: Baseline, week 8
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 329
participants | 309 | 288

27. Secondary Outcome: SBP Response 140 at Six Weeks
Description: SBP <140 mmHg or a reduction >=10 mmHg
Time Frame: Baseline, week 6
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 328
participants | 318 | 286

28. Secondary Outcome: SBP Response 140 at Four Weeks
Description: SBP <140 mmHg or a reduction >=10 mmHg
Time Frame: Baseline, week 4
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 329 | 326
participants | 309 | 274

29. Secondary Outcome: SBP Response 140 at Two Weeks
Description: SBP <140 mmHg or a reduction >=10 mmHg
Time Frame: Baseline, week 2
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 337 | 341
participants | 297 | 246

30. Secondary Outcome: SBP Response 140 at One Week
Description: SBP <140 mmHg or a reduction >=10 mmHg
Time Frame: Baseline, week 1
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 334 | 336
participants | 253 | 201

31. Secondary Outcome: SBP Response 130 at Eight Weeks
Description: SBP <130 mmHg or a reduction >=10 mmHg
Time Frame: Baseline, week 8
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 329
participants | 309 | 288

32. Secondary Outcome: SBP Response 130 at Six Weeks
Description: SBP <130 mmHg or a reduction >=10 mmHg
Time Frame: Baseline, week 6
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 328
participants | 318 | 286

33. Secondary Outcome: SBP Response 130 at Four Weeks
Description: SBP <130 mmHg or a reduction >=10 mmHg
Time Frame: Baseline, week 4
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 329 | 326
participants | 309 | 274

34. Secondary Outcome: SBP Response 130 at Two Weeks
Description: SBP <130 mmHg or a reduction >=10 mmHg
Time Frame: Baseline, week 2
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 337 | 341
participants | 297 | 246

35. Secondary Outcome: SBP Response 130 at One Week
Description: SBP <130 mmHg or a reduction >=10 mmHg
Time Frame: Baseline, week 1
Population: Treated set using LOCF
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 334 | 336
participants | 253 | 199

36. Secondary Outcome: DBP Response at Eight Weeks
Description: Mean seated DBP<80 mmHg or a reduction of <=10 mmHg
Time Frame: Week 8
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 329
participants | 253 | 214

37. Secondary Outcome: DBP Response at Six Weeks
Description: Mean seated DBP<80 mmHg or a reduction of <=10 mmHg
Time Frame: week 6
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 332 | 328
participants | 275 | 214

38. Secondary Outcome: DBP Response at Week Four
Description: Mean seated DBP <80 mmHg or a reduction of >=10 mmHg
Time Frame: Week 4
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 329 | 326
participants | 250 | 190

39. Secondary Outcome: DBP Response at Week Two
Description: Mean seated DBP <80 mmHg or a reduction of >=10 mmHg
Time Frame: Week 2
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 337 | 341
participants | 206 | 166

40. Secondary Outcome: DBP Response at Week One
Description: Mean seated DBP <80 mmHg or a reduction of >=10 mmHg
Time Frame: Week 1
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Telmisartan 80 mg + Amlodipine 5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 334 | 336
participants | 165 | 113

41. Secondary Outcome: Change From Baseline in Urine Albumin:Creatinine Ratio (UACR)
Description: Change from baseline in UACR (measured in spot urine) after eight weeks of treatment
Time Frame: 8 weeks
Population: Treated set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Number analyzed (Participants) | 334 | 333
ratio | -0.36 (0.79) | 0.04 (0.92)

ADVERSE EVENTS:
Arm/Group | Telmisartan 80 mg + Amlodipine 10 mg | Amlodipine 10 mg
Serious Adverse Events (participants affected / at risk) | 3/352 | 4/354
Other Adverse Events (participants affected / at risk) | 62/352 | 71/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 80 mg + Amlodipine 10 mg (N=352) | Amlodipine 10 mg (N=354)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Ulcer (General disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 80 mg + Amlodipine 10 mg (N=352) | Amlodipine 10 mg (N=354)
Oedema peripheral (General disorders) | 62 | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.